CLINICAL TRIAL: NCT06256510
Title: AN INTERVENTIONAL, PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD STUDY TO ESTIMATE THE EFFECT OF SINGLE AND MULTIPLE DOSES OF VEPDEGESTRANT (ARV-471, PF-07850327) ON THE PHARMACOKINETICS OF SINGLE DOSE MIDAZOLAM IN HEALTHY ADULT FEMALES OF NON-CHILDBEARING POTENTIAL.
Brief Title: A Study to Learn If the Study Medicine Called Vepdegestrant Changes How the Body Processes the Other Study Medicine Called Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C4891039; 2023-508518-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midazolam with and without Vepdegestrant (Experimental): Midazolam administered as a single dose in Period 1 Day 1, and Period 2 Day 1 and Day 15. Vepdegestrant administered once a day for 15 days in Period 2.
  Interventions: Drug: Midazolam; Drug: Vepdegestrant

INTERVENTIONS:
Drug: Midazolam — Participants will receive a single dose of Midazolam by mouth in Period 1 Day 1, and Period 2 Day 1 and Day 15
Drug: Vepdegestrant — Participants will receive Vepdegestrant by mouth once a day for 15 days in Period 2.
  Other Names: ARV-471; PF-07850327

SUMMARY:
The purpose of this study is to learn if the study medicine called Vepdegestrant changes how the body processes the other study medicine called Midazolam.

This study is seeking participants who:

* female who cannot have children.
* are 18 years or older.
* are overtly healthy as decided by medical tests.
* have a body mass index (BMI) of 16 to 32 kilogram per meter squared.
* have a total body weight of more than 45 kilograms (99 pounds).

All participants in this study will receive one dose of midazolam alone by mouth in Period 1. In Period 2, all participants will receive vepdegestrant by mouth once a day for 15 days. Participants will also receive one dose of midazolam by mouth on day 1 and day 15.

The levels of midazolam in Period 1 will be compared to the levels of midazolam in Period 2 Day 1 and Day 15 to decide if vepdegestrant affects how midazolam is processed differently in healthy adults.

The study duration is 22 days and includes two periods. Participants will stay in the clinical research unit through the end of period 2. A follow-up visit for each participant takes place at 28 to 35 days after taking the study medicine for the last time.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants of non-childbearing potential aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
2. Body mass index (BMI) of 16-32 kg/m2; and a total body weight >45 kg (99 lb).
3. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
4. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy)
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). Hepatitis B vaccination with an isolated positive hepatitis B surface antibody (HBsAb) result is allowed.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements, grapefruit/grapefruit containing products, and Seville orange/Seville orange containing products within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention. Refer to Section 6.9 Prior and Concomitant Therapy for additional details.

   * Moderate or strong CYP3A/P-gp inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
   * Moderate or strong CYP3A/P-gp inhibitors which are prohibited within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
4. Current use of any prohibited concomitant medication(s). Refer to Section 6.9 Prior and Concomitant Therapy.
5. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
6. A positive urine drug test or alcohol breath test at discretion of investigator. A single repeat for positive drug screen may be allowed.
7. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
8. Standard 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete left bundle branch block (LBBB), signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
9. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   • Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or Total Bilirubin Level ≥1.25 × upper limit of normal (ULN)
10. Renal impairment as defined by an estimated glomerular filtration rate (eGFR)<60 mL/min/1.73 m2. Based upon participant age at screening, eGFR is calculated using the recommended chronic kidney disease epidemiology (CKD-EPI) equations in Section 10.6.2 to determine eligibility and to provide a baseline to quantify any subsequent kidney safety events.
11. History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 4 or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
12. History of use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
13. History of hypersensitivity reactions to midazolam and vepdegestrant, or any of the formulation components of midazolam and vepdegestrant.
14. Unwilling or unable to comply with the criteria in the Section 5.3 of this protocol.
15. Investigator site staff directly involved in the conduct of the study and Investigator site staff's family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and site staff's, sponsor's and sponsor delegate's family members.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Midazolam when administered alone | Period 1 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
Cmax of Midazolam following multiple doses of Vepdegestrant | Period 2 - Day 15 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hour post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Midazolam when administered alone | Period 1 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
AUCinf of Midazolam following multiple doses of Vepdegestrant | Period 2 - Day 15 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hour post-dose

SECONDARY OUTCOMES:
Cmax of Midazolam following a single dose of Vepdegestrant | Period 2 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
AUCinf of Midazolam following a single dose of Vepdegestrant | Period 2 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to Period 2 Day 20
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Period 2 Day 20
Number of Participants With Electrocardiogram (ECG) Abnormalities | Baseline up to Period 2 Day 20
Number of Participants With Abnormalities in Physical Examinations | Baseline up to Period 2 Day 20
Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration (AUClast) of Midazolam when administered alone | Period 1 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
AUClast of Midazolam following multiple doses of Vepdegestrant | Period 2 - Day 15 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hour post-dose
AUClast of Midazolam following a slinge dose of Vepdegestrant | Period 2 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
Time for Cmax (Tmax) of Midazolam when administered alone | Period 1 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
Tmax of Midazolam following multiple doses of Vepdegestrant | Period 2 - Day 15 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hour post-dose
Tmax of Midazolam following a slinge dose of Vepdegestrant | Period 2 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
Apparent clearance (CL/F) of Midazolam when administered alone | Period 1 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
CL/F of Midazolam following multiple doses of Vepdegestrant | Period 2 - Day 15 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hour post-dose
CL/F of Midazolam following a slinge dose of Vepdegestrant | Period 2 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
Apparent volume of distribution (Vz/F) of Midazolam when administered alone | Period 1 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose
Vz/F of Midazolam following multiple doses of Vepdegestrant | Period 2 - Day 15 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hour post-dose
Vz/F of Midazolam following a slinge dose of Vepdegestrant | Period 2 - Day 1 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891039